CLINICAL TRIAL: NCT02107937
Title: A Randomized, Open-label, Three-arm, Multi-center Phase II Trial of Addition of DCVAC/OvCa to First Line Standard Chemotherapy in Women With Newly Diagnosed Epithelial Ovarian Carcinoma
Brief Title: Phase II Study DCVAC/OvCa Added to First Line Carboplatin and Paclitaxel Newly Diagnosed Epithelial Ovarian Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SOTIO a.s. (Industry)
Responsible Party: Sponsor
Organization: Sotio Biotech Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOV01; 2013-001322-26 (EudraCT Number)
Record Dates: First submitted 2014-04-04; First posted 2014-04-08 (Estimated); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Ovarian Neoplasms; Ovarian Epithelial Cancer
Keywords: serous; endometrioid; mucinous; epithelial ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Standard of Care; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- DCVAC/OvCa with Standard of Care (Experimental): DCVAC/OvCa in parallel with chemotherapy (Standard of Care)
  Interventions: Biological: DCVAC/OvCa with Standard of Care
- DCVAC/OvCa sequentially chemotherapy (Experimental): DCVAC/OvCa sequentially after chemotherapy
  Interventions: Biological: DCVAC/OvCa sequentially chemotherapy
- Standart of Care (Active Comparator): Carboplatin and Paclitaxel is Standard of Care First Line Chemotherapy
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Biological: DCVAC/OvCa with Standard of Care — DCVAC/OvCa is the experimental therapy added on to Carboplatin and Paclitaxel
  Other Names: Carboplatin; Paclitaxel
  Arms: DCVAC/OvCa with Standard of Care
Biological: DCVAC/OvCa sequentially chemotherapy — DCVAC/OvCa added sequentially after Carboplatin and Paclitaxel
  Other Names: Carboplatin; Paclitaxel
  Arms: DCVAC/OvCa sequentially chemotherapy
Drug: Standard of Care — Carboplatin and Paclitaxel is Standard of Care First Line Chemotherapy
  Other Names: Carboplatin; Paclitaxel
  Arms: Standart of Care

SUMMARY:
The purpose of this study is to determine whether DCVAC/OvCa added to chemotherapy (carboplatin plus paclitaxel as first line chemotherapy) may result in prolongation of progression free survival (PFS).

DETAILED DESCRIPTION:
The purpose of this study is to determine whether DCVAC/OvCa added to Standard of Care chemotherapy (carboplatin plus paclitaxel as first line chemotherapy) may result in prolongation of progression free survival (PFS).

ELIGIBILITY:
Inclusion Criteria:

* Female aged ≥18 years
* Patients with newly diagnosed, histologically confirmed, International Federation of Gynecology and Obstetrics (FIGO) stage III epithelial ovarian, primary peritoneal or fallopian tube carcinoma (serous, endometrioid or mucinous) who have undergone initial surgery up to 3 weeks before randomization and are selected to receive first line Standard of Care chemotherapy (optional prolongation to 6 weeks after surgery)
* Optimally debulked (zero residuum) or maximal residuum <1cm
* Eastern Cooperative Oncology Group (ECOG) Performance status 0,1,2

Exclusion Criteria:

* FIGO I,II,IV epithelial ovarian cancer
* FIGO III clear cells epithelial ovarian cancer
* Non-epithelial ovarian cancer (OvCa), borderline tumors (tumors of low malignant potential)
* Post-surgery residual disease with lesion(s) >1cm
* Prior or current systemic anti-cancer therapy for ovarian cancer [for example chemotherapy, monoclonal antibody therapy (bevacizumab), tyrosine kinase inhibitor therapy, vascular endothelial growth factor (VEGF) therapy or hormonal therapy]
* Previous or concurrent radiotherapy to the abdomen and pelvis
* Malignancy other than epithelial ovarian cancer, except those that have been in clinical remission (CR) for a minimum of 3 years, and except carcinoma in-situ of the cervix or non-melanoma skin carcinomas
* Patient co-morbidities:Human immunodeficiency virus (HIV) positive, human T-lymphotropic virus (HTLV) positive, Active hepatitis B (HBV), active hepatitis C (HCV), active syphilis
* Evidence of active bacterial, viral or fungal infection requiring systemic treatment
* Clinically significant cardiovascular disease including:

Symptomatic congestive heart failure Unstable angina pectoris Serious cardiac arrhythmia requiring medication Uncontrolled hypertension Myocardial infarction or ventricular arrhythmia or stroke within a 6 month period before inclusion, ejection fraction (EF) < 40 percent or serious cardiac conduction system disorders, if a pacemaker is not present

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2020-11 (Actual); Study Completion 2021-11 (Actual)

PRIMARY OUTCOMES:
Overall progression free survival (PFS) | 104 weeks

SECONDARY OUTCOMES:
Proportion of patients in remission after first line chemotherapy at 6 months | 0,10, 18, 30, 42 weeks
Proportion of patients in remission after first line chemotherapy at 12 months | 0,10, 18, 30, 42, 54, 68, 80, 92, 104 weeks
Biological progression free interval | 0,10, 18, 30, 42, 54, 68, 80, 92, 104 weeks
Immunological Response | 0, 6, 9, 12, 15, 18, 24, 30, 36, 42, 48, 54, 60 weeks
Proportion of patients requiring 2nd line chemotherapy | 0, 4, 6, 7, 9, 10, 12, 13, 15, 16, 18, 21, 24, 27, 30, 36, 42, 48, 54, 60, 64, 68, 74, 80, 86, 92, 98, 104 weeks
Frequency of Adverse Events | 0, 4, 6, 7, 9, 10, 12, 13, 15, 16, 18, 21, 24, 27, 30, 36, 42, 48, 54, 60, 64, 68, 74, 80, 86, 92, 98, 104 weeks
Time to 50 percent survival | 0, 4, 6, 7, 9, 10, 12, 13, 15, 16, 18, 21, 24, 27, 30, 36, 42, 48, 54, 60, 64, 68, 74, 80, 86, 92, 98, 104 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Harald Fricke, MD, PhD, Study Director — SOTIO a.s.
Locations (10):
- Czechia (8):
  - Brno
  - České Budějovice
  - Hradec Králové
  - Nový Jičín
  - Olomouc
  - Ostrava
  - Pilsen
  - Prague
- Poland (2):
  - Bialystok
  - Lublin

IPD SHARING:
Plan to Share IPD: Yes
EMA website

REFERENCES:
- [Derived] Hensler M, Rakova J, Kasikova L, Lanickova T, Pasulka J, Holicek P, Hraska M, Hrnciarova T, Kadlecova P, Schoenenberger A, Sochorova K, Rozkova D, Sojka L, Drozenova J, Laco J, Horvath R, Podrazil M, Hongyan G, Brtnicky T, Halaska MJ, Rob L, Ryska A, Coosemans A, Vergote I, Garg AD, Cibula D, Bartunkova J, Spisek R, Fucikova J. Peripheral gene signatures reveal distinct cancer patient immunotypes with therapeutic implications for autologous DC-based vaccines. Oncoimmunology. 2022 Jul 22;11(1):2101596. doi: 10.1080/2162402X.2022.2101596. eCollection 2022. PMID 35898703
- [Derived] Fucikova J, Hensler M, Kasikova L, Lanickova T, Pasulka J, Rakova J, Drozenova J, Fredriksen T, Hraska M, Hrnciarova T, Sochorova K, Rozkova D, Sojka L, Dundr P, Laco J, Brtnicky T, Praznovec I, Halaska MJ, Rob L, Ryska A, Coosemans A, Vergote I, Cibula D, Bartunkova J, Galon J, Galluzzi L, Spisek R. An Autologous Dendritic Cell Vaccine Promotes Anticancer Immunity in Patients with Ovarian Cancer with Low Mutational Burden and Cold Tumors. Clin Cancer Res. 2022 Jul 15;28(14):3053-3065. doi: 10.1158/1078-0432.CCR-21-4413. PMID 35536547
- [Derived] Rob L, Cibula D, Knapp P, Mallmann P, Klat J, Minar L, Bartos P, Chovanec J, Valha P, Pluta M, Novotny Z, Spacek J, Melichar B, Kieszko D, Fucikova J, Hrnciarova T, Korolkiewicz RP, Hraska M, Bartunkova J, Spisek R. Safety and efficacy of dendritic cell-based immunotherapy DCVAC/OvCa added to first-line chemotherapy (carboplatin plus paclitaxel) for epithelial ovarian cancer: a phase 2, open-label, multicenter, randomized trial. J Immunother Cancer. 2022 Jan;10(1):e003190. doi: 10.1136/jitc-2021-003190. PMID 34992091